CLINICAL TRIAL: NCT05501301
Title: Immune Tolerance After Pediatric Liver transplantation-a Cohort Study
Brief Title: Immune Tolerance After Pediatric Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Liu Yuan, Assistant professor, RenJi Hospital
Other Study IDs: IIT-2022-0004
Record Dates: First submitted 2022-08-07; First posted 2022-08-15 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Immune Tolerance; Liver Transplant; Complications
Keywords: immune tolerance, pediatric liver transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The peripheral blood samples and liver biopsy will be stored during study. Blood samples will be used for blood tests including liver function, IS level and immunological factors. Liver biopsy will be used for pathological evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immune tolerance cohort: Patients that are enrolled into this cohort will receive IS minimization if virus infection or side effects of IS was found. The strategy of IS minimization will follow the "Clinical guidelines for pediatric liver transplantation in China(2015)". Blood test and liver biopsy will be conducted to monitor liver function and intrahepatic pathological conditions. If IS is ceased for more than one year without liver dysfunction or signs of acute rejection in liver biopsy, immune tolerance was considered reached.
  Interventions: Other: IS weaning off

INTERVENTIONS:
Other: IS weaning off — IS weaning off will be conducted in recipients with chronic virus infection or side effects of IS

SUMMARY:
Immunosuppressive (IS) agents are effective treatment to avoid acute or chronic rejection after pediatric liver transplantation. However, long-term side effect of IS intaking, like infection, kidney dysfunction, metabolic disorders and developmental retardation, should be aware, especially in pediatric recipients. Spontaneous immune tolerance is defined as recipients who cease to taking IS agents due to multiple reasons and the liver function maintained normal. However, the real ratio and safety of immune tolerance in pediatric liver transplantation recipients are rarely known. We would like to investigate the ratio and safety of spontaneous immune tolerance in pediatric liver transplantation recipients during long-term follow-up by constructing an immune tolerance cohort. In this cohort, long-term pediatric liver transplantation recipients with normal liver function and taking monotherapy of IS would be involved. The IS strategy would be monitored and adjusted according to the "Clinical guidelines for pediatric liver transplantation in China(2015)". For recipients suffering refractory virus infection, such as EBV or CMV infection, IS will be minimized to assist the clearance of virus until IS was weaned off. Since most of pediatric liver transplantation recipients may encounter chronic EBV or CMV infection within one year after transplantation, they may need IS minimization during follow-up. During the process of IS weaning off, liver function, immunological status and intrahepatic pathology will be closely monitored. If acute rejection or other complications were found, increase of IS dosage or other related treatments will be applied. Immune tolerance is defined as liver function and intrahepatic pathology maintain normal for more than one year after stop taking IS. At the end of study, the ratio of immune tolerance, acute rejection and all types of complications will be assessed.

DETAILED DESCRIPTION:
Background: Immune tolerance after liver transplantation is defined as the status that recipients no longer taking any immunosuppressive agents with normal liver function and intrahepatic pathology. For pediatric liver transplantation recipients, immune tolerance is easier to reach than adult liver transplantation recipients. It is reported that spontaneous immune tolerance ratio in pediatric liver transplantation recipients is between 15%-60%, varying among different centers. Some recipients could develop into spontaneous immune tolerance due to refractory infections or side effects of IS. Some recipients could also reach immune tolerance by gradually weaning off the IS if liver function maintained normal and stable in the long-term follow-up. What's more, immune tolerance could reduce the long-term side effects of IS in pediatric recipients. However, how the immune status was modulated, or which factors contribute to the development of immune tolerance is unknown. Besides, the long-term safety of immune tolerance also needs more research. This study is designed to figure out the ratio and safety of immune tolerance in pediatric liver transplantation recipients.

Assessment before enrollment: In this study, enrolled population should have received living donor liver transplantation (LDLT) in Ren Ji Hospital affiliated to Shanghai Jiao Tong University School of Medicine for more than one year and liver function maintains stable and normal for more than 3 months. No severe complication including vessel complications, biliary complications or renal dysfunction should occur before enrollment. Liver biopsy should indicate no signs of acute rejection or chronic rejection, and no obvious fibrosis (Ishak<2).

Protocol after enrollment: After enrollment, the recipients will be evaluated for virus infection and side effects of IS. For patients with refractory EBV or CMV infections, or obvious side effects of IS, IS minimization should be applied. The dosage of IS will be weaned off as the 3/4 dosage of last dosage every 4 weeks. During the process of weaning off, liver function will be monitored every two weeks and liver biopsy should be conducted every six months. If liver dysfunction or acute rejection is detected during follow-up, steroid bolus and increased IS will be applied. For patients who have stop taking any IS, liver biopsy will be conducted to exclude potential liver injury in liver biopsy. For patients who have stop taking IS for more than one year with normal liver function and liver pathology, immune tolerance is considered as reached. At the endpoint of study, the ratio of immune tolerance, ratio of acute rejection and safety of immune tolerance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age at liver transplantation: 4 months to 18 years;
2. Original disease before liver transplantation: End-stage liver diseases including cholestatic diseases or metabolic diseases;
3. Type of liver transplantation: living donor liver transplantation, with donors of recipient's parents
4. Follow-up time after liver transplantation: more than one year
5. Liver function: liver function maintains normal and stable 3 months before enrollment
6. IS strategy: monotherapy of IS (FK or cyclosporine) or no longer taking any IS
7. Liver biopsy: No signs of acute rejection or chronic rejection, and no obvious fibrosis (Ishak<2)
8. Written consents are required

Exclusion Criteria:

1. Original disease before liver transplantation: Tumor, hepatitis virus infection, autoimmune hepatitis, liver failure, secondary liver transplantation
2. Type of liver transplantation: ABO incompatible liver transplantation, donors are not recipient's parents or multiple organ transplantation
3. Hepatitis virus infection during follow-up
4. Severe compilations, including bleeding complication, biliary complication, vessel complication or renal dysfunction -

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population is pediatric liver transplantation recipient that received living donor liver transplantation (LDLT) in Ren Ji Hospital affiliated to Shanghai Jiao Tong University School of Medicine. The enrolled recipients should have received LDLT for more than one year and liver function maintains stable and normal for more than 3 months. No severe complication including vessel complications, biliary complications or renal dysfunction should occur before enrollment. As for most recipient, monotherapy of IS will be applied three months after transplantation, so the enrolled recipients should taking only one type of IS. Since most of pediatric liver transplantation recipients may encounter chronic EBV or CMV infection with one year after transplantation, they may need IS minimization during follow-up. For those patients, IS weaning off will be applied. During the process of IS weaning off, liver function, immunological status and intrahepatic pathology will be closely monitored.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of immune tolerance | One year after withdraw of IS
  The ratio of spontaneous immune tolerance in pediatric liver transplantation recipients, which is free of IS for more than one year with normal liver function

SECONDARY OUTCOMES:
Ratio of acute rejection | 6 months, 1 year, 2 years and 3 years after enrolled into the study
  The ratio of acute rejection that happens in recipients during the process of IS minimization

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xia, MD, Study Director — Ren Ji Hospital affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ren Ji Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang B, Zhou A, Wu Y, Pan Q, Wei X, Gao Y, Xiao W, Jin J, Zhou T, Luo Y, Zhan Z, Liu Y, Gao W, Liu Y, Xia Q. Establishment and validation of a predictive model of immune tolerance after pediatric liver transplantation: a multicenter cohort study. Int J Surg. 2024 Sep 1;110(9):5615-5626. doi: 10.1097/JS9.0000000000001671. PMID 38833360